CLINICAL TRIAL: NCT05599789
Title: A Phase 2 Study of Pembrolizumab in Combination With Plinabulin and Docetaxel in Previously Treated Patients With Metastatic Non-Small Cell Lung Cancer and Progressive Disease (PD) After Immunotherapy (Anti-PD-1/PD-L1 Inhibitor) Alone or in Combination With Platinum-doublet Chemotherapy (KeyPemls-004)
Brief Title: Pembrolizumab in Combination With Plinabulin and Docetaxel For Metastatic NSCLC After ICIs (KeyPemls-004)
Acronym: KeyPemls-004
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: BeyondSpring Pharmaceuticals Inc. (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Wang mengzhao, Chief Director of Department of Respiratory and Critical Care Medicine, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K2506; BPI-2358-303 (Other: Beyondspring); MISP100168 (Other: MSD)
Record Dates: First submitted 2022-10-26; First posted 2022-10-31 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2024-03

CONDITIONS: Non Small Cell Lung Cancer Metastatic
Keywords: Carcinoma, Non-Small-Cell Lung; Pembrolizumab; Plinabulin; Docetaxel
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; NPI 2358; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pembrolizumab in Combination with Plinabulin and Docetaxel (Experimental): Pembrolizumab in Combination with Plinabulin and Docetaxel
  Interventions: Drug: Pembrolizumab in Combination with Plinabulin and Docetaxel

INTERVENTIONS:
Drug: Pembrolizumab in Combination with Plinabulin and Docetaxel — Pembrolizumab 200 mg Q3W IV infusion Day 1 of each 3-week cycle; Plinabulin 30 mg/m2 Q3W IV infusion Days 1 of each 3-week cycle; Docetaxel 75 mg/m² Q3W IV infusion Day 1 of each 3-week cycle.

SUMMARY:
A Phase 2 Study of Pembrolizumab in Combination with Plinabulin and Docetaxel in previously treated Patients with Metastatic Non-Small Cell Lung Cancer and progressive disease (PD) after immunotherapy (Anti-PD-1/PD-L1 inhibitor) alone or in combination with Platinum-doublet Chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female participants who are at least 18 years of age on the day of signing informed consent histologically confirmed diagnosis of metastatic squamous or non-squamous NSCLC (AJCC Staging Manual, version 8) will be enrolled in this study.
2. Male participants:

   A male participant must agree to use a contraception as detailed in Appendix 3 of this protocol during the treatment period and for at least 180 days after the last dose of study treatment and refrain from donating sperm during this period.
3. A female participant is eligible to participate if she is not pregnant (see Appendix 3), not breastfeeding, and at least one of the following conditions applies:

   1. Not a woman of childbearing potential (WOCBP) as defined in Appendix 3 OR
   2. A WOCBP who agrees to follow the contraceptive guidance in Appendix 3 during the treatment period and for at least 180 days after the last dose of study treatment.
   3. Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours prior to the start of study drug.
4. Participants must have progressed on treatment with an anti-PD-1/L1 mAb administered either as monotherapy or in combination with platinum-doublet chemotherapy.

   PD-1 treatment progression is defined by meeting all of the following criteria:
   1. Has received at least 2 doses of an approved anti-PD-1/L1 mAb.
   2. Has demonstrated disease progression after anti-PD-1/L1 as defined by RECIST v1.1.
   3. Progressive disease has been documented within 12 weeks from the last dose of anti-PD-1/L1 mAb.

      Once disease progression is confirmed, the initial date of disease progression documentation will be considered the date of disease progression.
   4. Progression-free survival of ICIs treatment at least 6 months： PD after platinum doublet chemotherapy AND immunotherapy either sequentially or concomitantly for advanced NSCLC with negative driver gene mutations.

   If subjects have disease progression within six months of the last dose of chemotherapy for neoadjuvant/adjuvant ICIs in combination with platinum-doublet chemotherapy for resectable NSCLC, the ICIs combination treatment can be defined as first-line treatment.

   For unresectable stage III NSCLC subjects who received CCRT followed by ICI as maintain treatment has disease progression within 1 year of the last dose of chemotherapy, the ICIs treatments can be defined as first-line treatment.
5. Have confirmation that EGFR-, ALK-, or ROS1-directed therapy is not indicated as primary therapy
6. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
7. Have measurable disease based on RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
8. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days before the first dose of the study intervention.
9. Have adequate organ function as defined in the following table. Specimens must be collected within 10 days before the start of the study intervention.
10. Have a life expectancy of at least 3 months.

Exclusion Criteria:

1. Has received docetaxel or Plinabulin as monotherapy or in combination with other therapies.
2. Has received other antitumor regimens before the initiation of the study regimen for those who had disease progression after prior ICI therapy.
3. Currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention.
4. Participants must have recovered from all AEs due to previous therapies to Grade 1 or less (except alopecia). Participants with ≤Grade 2 neuropathy may be eligible. Participants with endocrine-related AEs Grade ≤2 requiring treatment or hormone replacement may be eligible.
5. Major surgery, open biopsy, or obvious trauma within 4 weeks before enrollment.
6. Has received prior radiotherapy within 2 weeks before the start of study intervention or has received lung radiation therapy >30 Gy within 6 months before the first dose of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
7. Has received a live vaccine or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines is allowed. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
8. History of hemorrhagic diarrhea, inflammatory bowel disease or active uncontrolled peptic ulcer disease. (Concomitant therapy with ranitidine or its equivalent and/or omeprazole or its equivalent is acceptable). History of ileus or other significant gastrointestinal disorder known to predispose to ileus or chronic bowel hypomotility.
9. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
10. Known additional malignancy that is progressing or has required active treatment within the past 3 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ, excluding carcinoma in situ of the bladder, that have undergone potentially curative therapy are not excluded.
11. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression, clinically stable and without requirement of steroid treatment for at least 14 days prior to the first dose of study intervention.
12. Has severe hypersensitivity (≥Grade 3) to pembrolizumab/ Plinabulin/Docetaxel and/or any of its excipients.
13. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease-modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
14. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
15. Has an active infection requiring systemic therapy.
16. Has a known history of Human Immunodeficiency Virus (HIV) infection. Note: No HIV testing is required unless mandated by the local health authority.
17. Concurrent active Hepatitis B (defined as HBsAg positive and/or detectable HBV DNA) and Hepatitis C virus (defined as anti-HCV Ab positive and detectable HCV RNA) infection.

    Note: Hepatitis B and C screening tests are not required unless:

    Known history of HBV and HCV infection： As mandated by the local health authority.
18. Has known history of active TB (Bacillus Tuberculosis).
19. Any medical conditions that in the Investigator's opinion, would impose excessive risk to the patient. Examples of such conditions include uncontrolled diabetes, infection requiring parenteral anti-infective treatment, liver failure, any altered mental status or any psychiatric condition that would interfere with the understanding of the ICF. Has a history or current evidence of any condition, therapy, or laboratory abnormality or other circumstance that might confound the results of the study, interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator.
20. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
21. Pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 180 days after the last dose of trial treatment.
22. Has had an allogeneic tissue/solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-01-21 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR, objective response rate | through study completion, an average of 1 year
  the proportion of participants who have achieved a confirmed complete response (CR) or partial response (PR), which is assessed according to RECIST 1.1 criteria.

SECONDARY OUTCOMES:
PFS, progression-free survival | through study completion, an average of 1 year
  the time from treatment to the first documented progressive disease (PD) or death due to any cause, whichever occurs first.

OTHER OUTCOMES:
OS, overall survival | through study completion, an average of 1 year
  the time from allocation to the date of death due to any cause.
DOR, duration of response | through study completion, an average of 1 year
  the time from the first documented evidence of CR or PR until PD or death due to any cause, whichever occurs first, in participants demonstrating CR or PR
Adverse events (AEs) | through study completion, an average of 1 year
  Safety endpoints

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Respiratory and Critical Care Medicine, Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No